CLINICAL TRIAL: NCT02688361
Title: A Randomized, Open-Label, Two-Period, Crossover Bioequivalence Study in Healthy Adult Subjects After Single Oral Dosing of a NCH-GSK Acetylcysteine 2% Oral Solution Versus a Reference Fluimucil® Acetylcysteine 2% Oral Solution
Brief Title: A Bioequivalence Study of an Acetylcysteine 2% Oral Solution Versus a Reference Fluimucil 2% Oral Solution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 205033
Record Dates: First submitted 2016-02-18; First posted 2016-02-23 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2018-12

CONDITIONS: Infections, Respiratory Tract
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Acetylcysteine; Solutions

ARMS (2):
- Fluimucil® (reference) then Acetylcysteine (test) 2% solution (Experimental): Participants will be orally administered with 10ml of 2% oral solution of Fluimucil® (reference) following a wash out period of at least a week then administration of by 10ml of 2% oral solution of Acetylcysteine (test).
  Interventions: Drug: Fluimucil® 2% solution
- Acetylcysteine (test) 2% solution then Fluimucil® (reference) (Experimental): Participants will be orally administered with 10ml of 2% oral solution of Acetylcysteine (test) following a wash out period of at least a week then administration of by 10ml of 2% oral solution of Fluimucil® (reference).
  Interventions: Drug: Acetylcysteine 2% solution

INTERVENTIONS:
Drug: Fluimucil® 2% solution — Participants will be orally administered with 10ml of 2% oral solution of Fluimucil® (reference).
  Arms: Fluimucil® (reference) then Acetylcysteine (test) 2% solution
Drug: Acetylcysteine 2% solution — Participants will be orally administered with 10ml of 2% oral solution of Acetylcysteine (test)
  Arms: Acetylcysteine (test) 2% solution then Fluimucil® (reference)

SUMMARY:
This is an open-label, randomized, single-center, 2-period, 2-sequence, single-dose crossover design study in adult male and female healthy participants. Eligible participants will receive either treatment A (reference): Fluimucil® Acetylcysteine 2% oral solution, 200 mg N- acetylcysteine (NAC) in 10 mL dose, or treatment B (test): Acetylcysteine 2% oral solution, 200 mg NAC in 10 mL dose. Blood sampling will be collected pre-dose and up to 48 hours in each period. After completion of the second study period (i.e. last pharmacokinetic (PK) sample on Day 3 of Period 2) participants will be discharged from the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Participants must understand and provide written informed consent before any assessment is performed, understand the study procedures, and be willing to complete the required assessments.
* Male and female participants of any ethnic origin between 18 and 45 years of age. Body Mass Index (BMI) of 18.5 to 30 kg/m2, inclusive. Minimal body weight of 50 kg, inclusive.
* Normal vital signs as follows: Oral body temperature between 35.0 and 37.5 ºC inclusive; Sitting systolic blood pressure between 90 and 140 mmHg inclusive; Sitting diastolic blood pressure between 55 and 90 mmHg inclusive; Sitting pulse rate between 50 and 100 bpm inclusive.
* In general, good physical health, as judged by the Investigator and determined by medical/surgical history, physical examination, electrocardiogram (ECG, 12-lead) and clinical laboratory (clinical chemistry and hematology) findings.

Exclusion Criteria:

* Use of other investigational drugs within 3 months or 10 half-lives of enrollment, whichever is longer.
* History of or known hypersensitivity to any of the study drugs, excipients or to drugs of similar chemical or pharmacological classes.
* Diagnosis of long QT syndrome or QTc (Fridericia preferred, but Bazett acceptable) ≥ 450 msec for males and ≥ 470 msec for females at screening.
* History of malignancy or neoplastic disease of any organ system (except for localized basal cell skin carcinoma), treated or untreated, within the past 5 years prior to screening, regardless of whether there is evidence of local recurrence or metastases.
* Pregnant, Women of child-bearing potential or breastfeeding women.
* Any surgical or medical condition which may significantly alter the absorption, distribution, metabolism or excretion of any drug substance
* History (within 5 years prior to study start) of clinically significant gastritis, pyloric channel stenosis, peptic ulcer or duodenal ulceration, gastro-esophageal reflux, gastrointestinal bleeding, rectal bleeding or other clinically significant GI abnormalities.
* History (within 5 years prior to study start) of orthostatic hypotension, cardiovascular disease, stroke, transient ischemic attack, fainting or blackouts.
* Clinically relevant chronic or acute infectious illnesses or febrile infections within 2 weeks prior to start of the study.
* Newly occurred (within 2 weeks of screening visit) cutaneous and mucosal alterations.
* Participants with histamine intolerance.
* Positive results in any of the virology tests for Human Immunodeficiency Virus-Ab, Hepatitis C Antibody (HCV-Ab), Surface Antigen of the Hepatitis B Virus (HBsAg), and Hepatitis B Core Antibody (HBc-Ab).
* Any evidence of clinically significant cardiovascular, pulmonary, renal, hepatic, gastrointestinal, hematological, endocrinological, metabolic, autoimmune, neurological, psychiatric or other diseases at screening.
* Participant has used any medication (including over-the-counter medications) within 2 weeks before first scheduled study drug administration or within < 10 times the elimination halflife of the respective drug (whichever is longer), or is anticipated to require any concomitant medication during that period or at any time throughout the study.
* Participant reports consumption of any drug metabolizing enzyme (e.g. CYP3A4 or other cytochrome P450 enzymes) inducing or inhibiting aliments, beverages or food supplements within two weeks prior to the first scheduled study drug administration, or is anticipated to consume such products during that two-week period or at any time throughout the study.
* Any history of drug hypersensitivity, asthma, urticaria, or other significant allergic diathesis, illicit drug abuse.
* Participant shows evidence for current alcohol abuse or smoking.
* "Vulnerable" individuals.
* Participation in a previous clinical study with or without another investigational product and with ~470 ml blood drawn, or blood donation within the last 3 months prior to screening or previous enrollment into the current study.
* Any condition not identified in the protocol that, in the opinion of the Investigator, would confound the evaluation and interpretation of the study data or may put the participant at risk.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2016-04-13 (Actual); Study Completion 2016-04-13 (Actual)

PRIMARY OUTCOMES:
Area under the curve from time zero to last sampling time [AUC(0-last)] | 3 days
  AUC(0-last) of acetylcysteine will be calculated using trapezoidal rule. Blood samples will be taken pre-dose and upto 48 hours post-dose of administration of the reference/test product in each period.
Maximum Plasma Concentration (Cmax) | 3 days
  Cmax of acetylcysteine will be obtained graphically from the plasma concentration over time profile. Blood samples will be taken pre-dose and upto 48 hours post-dose of administration of the reference/test product in each period.

SECONDARY OUTCOMES:
Area under the curve from time zero to infinity [AUC(0-inf.)] | 3 days
  AUC(0-inf.) of acetylcysteine will be calculated using trapezoidal rule. Blood samples will be taken pre-dose and upto 48 hours post-dose of administration of the reference/test product in each period.
Time to reach maximum plasma concentration (Tmax) | 3 days
  Tmax of acetylcysteine will be obtained graphically from the plasma concentration over time profile. Blood samples will be taken pre-dose and upto 48 hours post-dose of administration of the reference/test product in each period.
Termination rate constant (Lambda_z) | 3 days
  Lambda_z will be computed as the slope of the regression line of ln (C(t)) on time.
Residual Area (RA) | 3 days
  RA will be calculated as percent extrapolated area (= (AUCinf - AUClast)/ AUCinf)*100%).
Elimination half life (t1/2) | 3 days
  T1/2 will be computed as T1/2 = 0.693/ λz

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Erfurt, Thuringia, Germany

REFERENCES:
- See also: Results for Study 205033 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/205033?search=study&study_ids=205033#rs